CLINICAL TRIAL: NCT05753826
Title: A Single-arm, Exploratory Study of Adebrelimab Combined With Fuzuloparib in the Treatment of Patients With Recurrent Platinum-resistant Ovarian Cancer
Brief Title: Adebrelimab Combined With Fuzuloparib in the Treatment of Patients With Recurrent Platinum-resistant Ovarian Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-OBU-FJ-OC-II-003
Record Dates: First submitted 2023-02-23; First posted 2023-03-03 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-10

CONDITIONS: Ovarian Neoplasms; Ovarian Diseases
MeSH Terms: conditions — Ovarian Neoplasms; Ovarian Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab Combined With Fuzuloparib (Experimental)
  Interventions: Drug: Adebrelimab; Drug: Fuzuloparib

INTERVENTIONS:
Drug: Adebrelimab — 20mg/kg，D1，q3W
Drug: Fuzuloparib — 100 mg bid

SUMMARY:
This is a single-arm, exploratory study. People with recurrent platinum-resistant ovarian cancer who have not received any previous systemic antitumor therapy for ovarian cancer were selected to evaluate the efficacy and safety of adebrelimab combined with fuzuloparib.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70;Female;
2. Pathologically (including histologically) confirmed epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer (hereinafter referred to as ovarian cancer), recurrence within less than 6 months after the last treatment with platinum-containing chemotherapy;
3. Patients have at least one target lesion with measurable dimensions according to RECIST1.1 criteria;
4. HRR gene mutation confirmed by testing tissue or blood samples;
5. ECOG PS 0-1;
6. Major organ functions are normal and meet the following criteria:(1) Blood routine inspection standards must meet: (no blood transfusion within 14 days)a.HB≥100g/L, b. WBC≥3×10^9/L c. ANC≥1.5×10^9/L, d.PLT≥100×10^9/L; (2) Biochemical examination must meet the following standards: a. BIL ≤1.5 times the upper limit of normal (ULN); b. ALT and AST≤2.5×ULN, ALT and AST≤5×ULN in patients with liver metastases; c. Serum Cr≤1.5×ULN
7. Activated partial thromboplastin time (APTT) ≤ 1.5 times ULN, prothrombin time (PT) ≤ 1.5 times ULN, international normalized ratio (INR) ≤ 1.5 times ULN, unless the patient is receiving anticoagulation, as long as PT or APTT is within the expected range of anticoagulant use;
8. No severe heart, lung, liver or kidney disorders;
9. Women of childbearing age must have a pregnancy test (serum) within 7 days prior to enrollment and have a negative result, and be willing to use appropriate methods of contraception during the trial period and 8 weeks after the last administration of the test drug;
10. Estimated survival≥ 12 weeks;
11. Sign a written informed consent form and be able to comply with the visitation and related procedures set out in the programme.

Exclusion Criteria:

1. Other clinical drug experiments in which other experimental research drugs are used concurrently with the study;
2. Patients with known hypersensitivity to fluzoparib or hypersensitivity to drug-active or inactive ingredients with a similar chemical structure to fluzoparib;
3. Patients with known hypersensitivity to adebrelimab or hypersensitivity to the active or inactive components of the drug having a similar chemical structure to adebrelimab;
4. Inability to swallow oral medications and any gastrointestinal disorders that may interfere with the absorption and metabolism of study medications, such as uncontrolled nausea and vomiting, gastrointestinal obstruction or malabsorption;
5. prior treatment with known or probable immune checkpoint inhibitors;
6. Have any active autoimmune disease or history of autoimmune disease (e.g., interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); Except vitiligo or recovered childhood asthma/allergies who do not require any intervention in adulthood; Autoimmune-mediated hypothyroidism treated with stable doses of thyroid-replacement hormones; Type I diabetes mellitus with a stable dose of insulin;
7. A history of immunodeficiency, including a positive HIV test, or other acquired or congenital immunodeficiency disorders, or a history of organ transplantation and allogeneic bone marrow transplantation;
8. With unstable systemic diseases, such as hypertension that cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥90 mmHg), severe arrhythmias, etc.;
9. Previous or current idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, organising pneumonia, drug-induced pneumonia, or active pneumonia on screening-phase CT;
10. There are cardiac clinical symptoms or diseases that are not well controlled, such as: (1) cardiac insufficiency above NYHA grade 2 (2) unstable angina (3) acute myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention (5) QTc>470ms;
11. Patients who are pregnant or breastfeeding, or who plan to become pregnant during study treatment;
12. The investigators considered it unsuitable for inclusion.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | 3 years
  ORR is determined using RECIST v1.1, Defined as the optimal overall response (CR or PR) at the time point assessed from enrollment to the end of neoadjuvant therapy

SECONDARY OUTCOMES:
Overall survival(OS) | 3 years
  Defined as the time from the enrollment to death from any cause
Progression free survival(PFS) | 3 years
  It is defined as the time from enrollment to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first.
Disease Control Rate(DCR) | 3 years
  DCR is determined using RECIST v1.1, Defined as the rate of disease control (CR or PR or SD) from enrollment to the end of neoadjuvant therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Sun, Doctor, Principal Investigator — Fujian Cancer Hospital
Locations (1):
- Fujian Cancer Hospital, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided